CLINICAL TRIAL: NCT06431672
Title: The Feasibility and Effects of Perinatal Interpersonal Psychotherapy Group for Distressed Women
Brief Title: Perinatal Interpersonal Psychotherapy Group for Distressed Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Peyling Shieh, Associate professor, Chung Shan Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOST 106-2410-H-040-004 -SSS; MOST 107-2410-H-040-005 -SSS (Other Grant/Funding Number: Ministry of Science and Technology, Taiwan)
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Depression, Postpartum; Social Adjustment
Keywords: feasibility; group psychotherapy; interpersonal psychotherapy; maternal depression; perinatal adjustment
MeSH Terms: conditions — Depression, Postpartum; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention was an eight-session P-IPTG, which consisted of four sessions in pregnancy and four in postpartum. All participants replied to the measures at four waves from baseline to one year postpartum. The outcome variables were within-group and between-group changes in depression, social support, dyadic adjustment, interpersonal relationship satisfaction, and mother-infant bonding.
  Interventions: Other: interpersonal group psychotherapy
- control group (No Intervention): The participants of control group reply questionnaires for four times.

INTERVENTIONS:
Other: interpersonal group psychotherapy — Interpersonal psychotherapy (IPT) was developed by Stuart and O'Hara (1995). It addresses four domains of conflict. The intervention is an eight-session P-IPTG, which consisted of four sessions in pregnancy and four in postpartum.
  Arms: intervention group

SUMMARY:
This is the first perinatal interpersonal psychotherapy group (P-IPTG) implemented for distressed women from pregnancy to postpartum. The feasibility and effects of P-IPTG are explored.

DETAILED DESCRIPTION:
This is the first perinatal interpersonal psychotherapy group (P-IPTG) implemented for distressed women from pregnancy to postpartum. The feasibility and effects of P-IPTG are explored. The third-trimester women were recruited as intervention and control group participants by a quasi-experimental design.

ELIGIBILITY:
Inclusion Criteria:

* women in the third trimester of pregnancy, at least 20 years old, able to read and write in Chinese, and "depressed, anxious, or wishing to improve family relationships."

Exclusion Criteria:

* women with schizophrenia, substance use, or suicide risk.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women in pregnancy and postpartum
Enrollment: 258 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | the seventh to ninth month in pregnancy, four month postpartum, eight month postpartum,twelve month postpartum
  The Edinburgh Postnatal Depression Scale (EPDS, Cox et al., 1987) was used to assess depressive symptoms. It consists of ten Likert-type items with 0 to 3 points, with higher scores indicating more depressive symptoms over the past week. Following the previous study (Su et al., 2007), we used higher than 12 to define participants with significant depressive tendencies.
Dyadic Adjustment Scale | the seventh to ninth month in pregnancy, four month postpartum, eight month postpartum,twelve month postpartum
  The Dyadic Adjustment Scale (DAS, Spanier, 1976) assessed women's perceived quality of either married or unmarried couple relationship. The scale consists of 32 items, primarily scored in a 6-point scale (27 items). It measures four factors: dyadic consensus, dyadic satisfaction, dyadic cohesion, and affectionate expression. Higher scores indicate better dyadic adjustment in respective aspects.
Social Network Interaction System Questionnaire (SNISQ, Lay & Liu, 1996) | the seventh to ninth month in pregnancy, four month postpartum, eight month postpartum,twelve month postpartum
  The Social Network Interaction System Questionnaire (SNISQ, Lay & Liu, 1996) was used to evaluate perceptions of social support from partners, original families, and in-laws. The SNISQ consists of nine Likert-type items with 1 to 4 points, with higher scores indicating better- perceived support from specific individuals.
Satisfaction with Interpersonal Relationships Scale (Chan et al., 2002) | the seventh to ninth month in pregnancy, four month postpartum, eight month postpartum,twelve month postpartum
  Chan et al. (2002) used the Satisfaction with Interpersonal Relationships Scale (SWIRS,) to assess women's satisfaction with their relationships with partners and mothers-in-law over the past few weeks. We expanded the scale to include ratings of relationships with fathers, mothers, and fathers-in-law, resulting in five items. The SWIRS is a Likert-type item with 1 to 7 points, with higher scores indicating greater satisfaction with the relationship.
Mother-Infant Bonding Inventory (Shieh et al., 2015) | the seventh to ninth month in pregnancy, four month postpartum, eight month postpartum,twelve month postpartum
  The Mother-Infant Bonding Inventory (MIBI, Shieh et al., 2015) assessed mothers' thoughts, feelings, and commitment toward their infants. The MIBI consists of 25 items scored on 1 to 6 points. Its four factors are proximity, parental adjustment, commitment, and confidence of reciprocity. Higher scores indicate good mother-infant bonding in specific aspects.

CONTACTS AND LOCATIONS:
Overall Officials: Peyling Shieh, Ph. D., Principal Investigator — Chung Shan Medical University, Taiwan
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
For confidentiality, we plan to share IPD with other researchers by contact.